CLINICAL TRIAL: NCT05568901
Title: Impact of Gun Lock Distribution on Firearm Securement After Emergent Mental Health Evaluation: A Randomized Controlled Trial
Brief Title: Randomized Trial to Improve Safe Firearm Storage
Acronym: FARTHER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Ohio Injury Prevention Partnership (Unknown); Whitney Strong Organization (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-0828
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Firearm Injury; Pediatric Emergency Medicine; Suicide and Self-harm; Mental Health Issue
Keywords: Suicide prevention; Pediatric; Firearm safety
MeSH Terms: conditions — Suicide; Self-Injurious Behavior; Suicide Prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LMC Alone (Active Comparator): Caregivers who received standardized lethal means counseling (LMC) from the study team as well as a 1-page handout summarizing the counseling recommendations
  Interventions: Behavioral: Lethal means counseling
- LMC + Gun Locks (Experimental): Caregivers who received standardized lethal means counseling (LMC) from the study team, 1-page handout summarizing the counseling recommendations, as well as the additional provision of 2 cable-style gun locks
  Interventions: Behavioral: Lethal means counseling; Behavioral: Provision of Cable-style gun locks

INTERVENTIONS:
Behavioral: Lethal means counseling — Lethal means counseling is a type of safety education that advises securement or removal of potentially hazardous household items such as medications, knives, and firearms. Counseling provided by study team was derived from the Suicide Prevention Resource Center's "Counseling on Access to Lethal Means" training module and the "Store It Safe" campaign from the Ohio Chapter of the American Academy of Pediatrics (AAP). Guidance focused on securement of dangerous items in the household, such as medications and firearms, with locking devices-or more preferably removing these items from the home, even if temporarily.
Behavioral: Provision of Cable-style gun locks — Caregivers were provided 2 (two) SnapSafe Cable Padlock (Item No. 75281), advised on how to use these devices to store firearms safely (including instructions from within the package of the provided gun locks) and were advised to store keys away from the firearm in a location that children would not have access
  Arms: LMC + Gun Locks

SUMMARY:
The goal of this clinical trial is to test the effect of providing gun locks to caregivers of children presenting to the emergency department for mental health concerns. The main question it aims to answer is:

• Does the provision of gun locks result in higher rates of securement of all household firearms? Participants will be randomized to receive either lethal means counseling (including summary handout) by study team with the provision of 2 cable-style gun locks or lethal means counseling by study team alone (without provision of gun locks).

Researchers will compare the lethal means counseling with 2 gun locks group to the lethal means counseling alone group to see if it affects self-reported securement of all household firearms, 4 weeks post emergency department encounter.

DETAILED DESCRIPTION:
Study Design and Population We conducted a single-center, prospective, randomized controlled trial with the emergency department of a free-standing tertiary care level-1 pediatric trauma center. Due to the nature of the study, investigators were not blinded to the interventions received by participants. This study was approved by the Cincinnati Children's Hospital Medical Center (CCHMC) Institutional Review Board. Study protocol, counseling handout, and surveys are available upon request to study team.

The study population consisted of firearm-owning caregivers of patients presenting to the PED for emergent MH evaluation. As only patients under the age of 18 can receive psychiatric care at our facility, all children of enrolled caregivers were less than 18 years of age.

Survey Development Survey content was derived from the expert opinion of PED physicians, injury prevention researchers, and psychiatry staff involved in the care of MH patients. Pre-counseling surveys contained questions regarding caregiver demographics as well as firearm and medication storage practices. Follow-up surveys repeated questions about storage behaviors with additional questions regarding how participants viewed PED-based counseling, use of the provided locks, removal of lethal means from the home, and the purchase of additional safety devices after PED encounter.

Counseling handouts and surveys were piloted for readability and content among 12 firearm-owning caregivers.17 Inclusion criteria revised to include all gun-owning caregivers rather than only those with unsafely stored weapons. Potential participants felt more comfortable relaying storage practices via anonymous survey as opposed to face-to-face with counselor during screening process. Content regarding another lethal mean, medication, was added to reduce perceived judgement surrounding firearm ownership.

Study Procedure All enrollment occurred within the primary PED of CCHMC between June 28, 2021 and February 10, 2022. Potential participants were identified by documented chief complaint of "Psychiatric Evaluation", which includes, but is not limited to, those presenting for: suicidal ideation/attempt, homicidal ideation/attempt, aggression, behavior change, and hallucinations. The Psychiatric Intake and Response Center (PIRC) team is made up of social workers and an attending psychiatrist that consult on all patients presenting to the PED for psychiatric evaluation. Caregivers who met inclusion criteria and received consultation by PIRC team were considered for enrollment. A convenience sample of caregivers were screened for enrollment by the study principal investigator (PI) or Clinical Research Coordinators (CRCs) specifically trained in study recruitment and lethal means counseling. CRCs were present in the PED 8am to 12pm on weekdays and 11am to 9pm on weekends. The PI aided in recruitment, as needed during high patient volumes.

Caregivers were approached for enrollment after patient had been evaluated by both emergency physicians and PIRC team. If more than one caregiver was present, one caregiver was chosen by the family for participation. Participants provided electronic consent prior to completing survey questions. Neither consent nor assent was required from patients as no protected health information was collected. Eligibility screening and safety counseling with caregiver occurred outside of patient room, physically distant from patient, in order to avoid raising awareness of firearms in the home. Baseline survey, detailing caregiver demographics as well as storage habits of medications and firearms, was completed prior to counseling.

Enrollment occurred in parallel with a 1:1 allocation ratio. Enrolled caregivers were randomized into one of two study arms based on date of enrollment. Participants enrolled on odd-numbered dates were allocated to the control group (LMC alone), while participants enrolled on even-numbered dates were allocated to the intervention group (LMC + 2 cable-style gun locks). Participants completed the electronic-based survey on a tablet with study team member present to clarify questions. The REDCap® application was used for data collection.

The control arm of the study received standardized LMC from the study PI or CRC as well as a 1-page handout summarizing the counseling recommendations. The intervention arm received the same counseling and handout with the additional provision of 2 cable-style gun locks. Counseling provided by study team was derived from the Suicide Prevention Resource Center's "Counseling on Access to Lethal Means" training module18 and the "Store It Safe" campaign19 from the Ohio Chapter of the American Academy of Pediatrics (AAP). Guidance focused on securement of dangerous items in the household, such as medications and firearms, with locking devices-or more preferably removing these items from the home, even if temporarily. Particular attention was given to the AAP's recommendations on safe storage of firearms, which states that all firearms should be kept locked, unloaded, with ammunition secured separately19. The cable locks were SnapSafe Cable Padlock (Item No. 75281). Cable locks were chosen as they have several advantages over other types of gun locks, including: (1) they are near-universally applicable to both handguns and long guns (2) cable locks are the least expensive type of gun locks, often costing 5-10x less than even the most basic gun safes/lockboxes (3) the possibility of unintentional discharge during securement process is much lower than that of devices such as a trigger locks and (4) even if a gun is kept loaded, a cable lock will prevent the firing pin from striking a bullet/shell. Caregivers were provided with instructions included within the package of the provided gun locks and advised to store keys away from the firearm in a location that children would not have access. All patients and caregivers received usual care from PIRC team which includes a standardized safety checklist and instructions on increased supervision of child. Counseling provided by study team members was supplementary to usual care.

A link to a follow-up survey was sent to participants 4 weeks after completion of baseline survey. This survey was distributed via text message using functionality within the REDCap® application and sent to the mobile phone of the participant completing the initial survey. If a participant did not complete the follow-up survey, reminders were sent at 3-day intervals up to 3 additional times. Participants received $10 gift cards upon completion of each survey.

Statistical Analysis A sample size of 200 patients was determined based on a 95% confidence interval with an 80% power to detect a 30% difference in primary outcome-based on described outcome differences in previous clinic-based trials.14 Sample size calculations accounted for an estimated 30% loss to follow-up based on prior survey-based projects within CCHMC PED.11 Wilcoxon rank sum and Fisher's exact tests were used to analyze differences between primary comparison groups at both baseline and follow-up, for continuous and categorical variables, respectively. Odds ratios and McNemar's test were used to compare baseline vs follow-up securement rates within and between study groups. Logistic regression-with adjustments for patient and caregiver age, gender and race-was used to compare change in proportion reporting firearm securement between study arms.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of pediatric patient presenting to the emergency department for mental health evaluation
* Caregiver endorses firearms within the home

Exclusion Criteria:

* Caregiver not present
* Caregiver is not able to complete survey in written English
* Caregiver unable to be approached due to unsafe conditions as determined by study team and behavioral safety specialists

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Firearm securement | 4 weeks post-encounter
  Self-reported securement of all household firearms with locking device

SECONDARY OUTCOMES:
Caregiver favorability | 4 weeks post-encounter
  Caregivers were asked their perceptions on the counseling they received from the choices: "Very Negatively, Somewhat Negatively, No opinion/Do not remember counseling, Somewhat Favorably, Very Favorably"
Medication securement | 4 weeks post-encounter
  Self-reported securement of all household medications with locking device
Firearm removal | 4 weeks post-encounter
  Self-reported removal of firearms from the home (permanent or temporary)
Medication removal | 4 weeks post-encounter
  Self-reported removal of medication from the home (permanent or temporary)
Additional devices | 4 weeks post-encounter
  Self-reported purchase of any additional safety devices (such as gun lock or lockbox)
Use of locks | 4 weeks post-encounter
  Self-reported use of 2 cable-style gun locks among those who received gun locks during counseling
Change in firearm securement | 4 weeks
  Change (pre vs post encounter) in proportion of households reporting all firearms secured
Change in medication securement | 4 weeks
  Change (pre vs post encounter) in proportion of households reporting all medications secured

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Web-based Injury Statistics Query and Reporting System (WISQARS). National Center for Health Statistics (NCHS). 2022. www.cdc.gov/injury/wisqars
- [Background] Miller M, Azrael D, Hemenway D. The epidemiology of case fatality rates for suicide in the northeast. Ann Emerg Med. 2004 Jun;43(6):723-30. doi: 10.1016/j.annemergmed.2004.01.018. PMID 15159703
- [Background] Grossman DC, Mueller BA, Riedy C, Dowd MD, Villaveces A, Prodzinski J, Nakagawara J, Howard J, Thiersch N, Harruff R. Gun storage practices and risk of youth suicide and unintentional firearm injuries. JAMA. 2005 Feb 9;293(6):707-14. doi: 10.1001/jama.293.6.707. PMID 15701912
- [Background] Beidas RS, Rivara F, Rowhani-Rahbar A. Safe Firearm Storage: A Call for Research Informed by Firearm Stakeholders. Pediatrics. 2020 Nov;146(5):e20200716. doi: 10.1542/peds.2020-0716. Epub 2020 Oct 9. No abstract available. PMID 33037120
- [Background] Azrael D, Cohen J, Salhi C, Miller M. Firearm Storage in Gun-Owning Households with Children: Results of a 2015 National Survey. J Urban Health. 2018 Jun;95(3):295-304. doi: 10.1007/s11524-018-0261-7. PMID 29748766
- [Background] Johnson RM, Barber C, Azrael D, Clark DE, Hemenway D. Who are the owners of firearms used in adolescent suicides? Suicide Life Threat Behav. 2010 Dec;40(6):609-11. doi: 10.1521/suli.2010.40.6.609. PMID 21198329
- [Background] Monuteaux MC, Azrael D, Miller M. Association of Increased Safe Household Firearm Storage With Firearm Suicide and Unintentional Death Among US Youths. JAMA Pediatr. 2019 Jul 1;173(7):657-662. doi: 10.1001/jamapediatrics.2019.1078. PMID 31081861
- [Background] Kalb LG, Stapp EK, Ballard ED, Holingue C, Keefer A, Riley A. Trends in Psychiatric Emergency Department Visits Among Youth and Young Adults in the US. Pediatrics. 2019 Apr;143(4):e20182192. doi: 10.1542/peds.2018-2192. Epub 2019 Mar 18. PMID 30886112
- [Background] Barkin SL, Finch SA, Ip EH, Scheindlin B, Craig JA, Steffes J, Weiley V, Slora E, Altman D, Wasserman RC. Is office-based counseling about media use, timeouts, and firearm storage effective? Results from a cluster-randomized, controlled trial. Pediatrics. 2008 Jul;122(1):e15-25. doi: 10.1542/peds.2007-2611. PMID 18595960
- [Background] Albright TL, Burge SK. Improving firearm storage habits: impact of brief office counseling by family physicians. J Am Board Fam Pract. 2003 Jan-Feb;16(1):40-6. doi: 10.3122/jabfm.16.1.40. PMID 12583649
- [Background] Gittelman MA, Pomerantz WJ, Laurence S. An emergency department intervention to increase booster seat use for lower socioeconomic families. Acad Emerg Med. 2006 Apr;13(4):396-400. doi: 10.1197/j.aem.2005.11.002. Epub 2006 Mar 10. PMID 16531596
- [Background] Runyan CW, Becker A, Brandspigel S, Barber C, Trudeau A, Novins D. Lethal Means Counseling for Parents of Youth Seeking Emergency Care for Suicidality. West J Emerg Med. 2016 Jan;17(1):8-14. doi: 10.5811/westjem.2015.11.28590. Epub 2016 Jan 12. PMID 26823923
- [Background] Uspal NG, Strelitz B, Cappetto K, Tsogoo A, Jensen J, Rutman LE, Schloredt K, Bradford MC, Bennett E, Paris CA. Impact of a Firearm Safety Device Distribution Intervention on Storage Practices After an Emergent Mental Health Visit. Acad Pediatr. 2021 Sep-Oct;21(7):1209-1217. doi: 10.1016/j.acap.2021.04.024. Epub 2021 May 1. PMID 33945885
- [Background] Carbone PS, Clemens CJ, Ball TM. Effectiveness of gun-safety counseling and a gun lock giveaway in a Hispanic community. Arch Pediatr Adolesc Med. 2005 Nov;159(11):1049-54. doi: 10.1001/archpedi.159.11.1049. PMID 16275796
- [Background] Posner JC, Hawkins LA, Garcia-Espana F, Durbin DR. A randomized, clinical trial of a home safety intervention based in an emergency department setting. Pediatrics. 2004 Jun;113(6):1603-8. doi: 10.1542/peds.113.6.1603. PMID 15173480
- [Background] Rowhani-Rahbar A, Simonetti JA, Rivara FP. Effectiveness of Interventions to Promote Safe Firearm Storage. Epidemiol Rev. 2016;38(1):111-24. doi: 10.1093/epirev/mxv006. Epub 2016 Jan 13. PMID 26769724
- [Background] Sheatsley PB. Handbook of Survey Research. In: Rossi PH, ed. Handbook of Survey Research. Academic Press; 1983:chap Chapter 6: Questionnaire Construction and Item Writing.
- [Background] Ruch DA, Steelesmith DL, Warner LA, Bridge JA, Campo JV, Fontanella CA. Health Services Use by Children in the Welfare System Who Died by Suicide. Pediatrics. 2021 Apr;147(4):e2020011585. doi: 10.1542/peds.2020-011585. Epub 2021 Mar 8. PMID 33685986
- [Background] Ketabchi B, Gittelman MA, Southworth H, Arnold MW, Denny SA, Pomerantz WJ. Attitudes and perceived barriers to firearm safety anticipatory guidance by pediatricians: a statewide perspective. Inj Epidemiol. 2021 Sep 13;8(Suppl 1):21. doi: 10.1186/s40621-021-00319-9. PMID 34517906
- [Derived] Ketabchi B, Gittelman MA, Zhang Y, Pomerantz WJ. Impact of cable lock distribution on firearm securement after emergent mental health evaluation: a randomized controlled trial. Inj Epidemiol. 2024 Nov 11;11(Suppl 1):63. doi: 10.1186/s40621-024-00541-1. PMID 39529188
- See also: Suicide prevention resource center's online "Counseling on access to lethal means" training module that was used to help develop lethal means counseling provided in the study — https://zerosuicidetraining.edc.org/enrol/index.php?id=20
- See also: Ohio Chapter of the American Academy of Pediatrics "Store it safe" campaign that was used to help develop lethal means counseling provided in the study — https://ohioaap.org/storeitsafe

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT05568901/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT05568901/ICF_001.pdf